CLINICAL TRIAL: NCT00669201
Title: Wrist Cartilage - High Resolution in Vivo MR T2 Mapping- a Feasibility Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Iris Eshed, MD, Sheba Medical Center
Other Study IDs: SHEBA-08-4912-IE-CTIL
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Osteoarthritis
Keywords: cartilage; osteoarthritis; T2 mapping; MRI; Wrist
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: healthy young volunteers Inclusion: age 18-40, Exclusion: wrist trauma/surgery
- 2: patients with know osteoarthritis wrist changes according to pre-existing x-rays No age limits
  exclusion: previous wrist surgery
- 3: Mixed group of 50 patients that perform routine MRI of the wrist for various indications

SUMMARY:
Purpose:Evaluate the feasibility of T2 cartilage mapping on MRI of the wrist and correlate with T2 mapping of knee cartilage.

Study protocol: Phase 1. 10 healthy volunteers, Phase 2. 10 volunteers with osteoarthritis of the wrist, Phase 3. 50 patients for studies for routine MR of the wrist.

MRI protocol: 3 T unit((Signa EXITE HDx),T1, T2 and T2 mapping sequences on axial and coronal orientation.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1. Age:18-40
* Phase 2: No age limit, known OA on pre-existing X-rays
* Phase 3: No age limit, routine MRI of the wrist

Exclusion Criteria:

* Phase 1, 2: wrist trauma/surgery
* All phases: any contraindication for MR: eg metals, claustrophobia, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers, volunteers with known osteoarthritis, routine MR population for wrist investigation
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2007-12

PRIMARY OUTCOMES:
wrist bone cartilage thickness can be measured and stratification can be observed on T2 mapping with correlation to T2 mapping of the knee cartilage | Within MRI completion (20 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Iris Eshed, MD, Principal Investigator — Sheba Medical Center
Locations (2):
- Israel (2):
  - Sheba Medical Center , Diagnostic Imaging Dept, Tel Litwinsky, Tel Hashomer
  - Sheba Medical Center, Diagnostic Imaging Dept, Tel Litwinsky, Tel Hashomer

REFERENCES:
- [Background] Glaser C. New techniques for cartilage imaging: T2 relaxation time and diffusion-weighted MR imaging. Radiol Clin North Am. 2005 Jul;43(4):641-53, vii. doi: 10.1016/j.rcl.2005.02.007. PMID 15893528
- [Background] Recht MP, Goodwin DW, Winalski CS, White LM. MRI of articular cartilage: revisiting current status and future directions. AJR Am J Roentgenol. 2005 Oct;185(4):899-914. doi: 10.2214/AJR.05.0099. PMID 16177408
- [Background] Mosher TJ, Dardzinski BJ, Smith MB. Human articular cartilage: influence of aging and early symptomatic degeneration on the spatial variation of T2--preliminary findings at 3 T. Radiology. 2000 Jan;214(1):259-66. doi: 10.1148/radiology.214.1.r00ja15259. PMID 10644134